CLINICAL TRIAL: NCT02265055
Title: Early Embryo Cleavage And Multiple Pregnancies After ICSI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, Obstetrics and Gynecology Department, faculty of medicine (Assiut), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: u12345
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

ARMS (2):
- transfer early cleavage embryos (EC) (Active Comparator): transfer early cleavage embryos
  Interventions: Procedure: transfer early cleavage embryos
- transfer non early cleavage embryo (NEC) (Active Comparator): transfer non early cleavage embryos
  Interventions: Procedure: transfer non early cleavage embryo

INTERVENTIONS:
Procedure: transfer early cleavage embryos — transfer early cleavage embryos
  Arms: transfer early cleavage embryos (EC)
Procedure: transfer non early cleavage embryo
  Arms: transfer non early cleavage embryo (NEC)

SUMMARY:
To observe whether Number of early cleavage embryos can be a predictor for multiple pregnancies after ICSI.

DETAILED DESCRIPTION:
A total of 193 infertile couples, attending the ART unit, International Islamic Center for Population Studies and Research (IICPSR), -Al- Azhar University in the period from December 2010 to September 2012, were included in this study.

The controlled ovarian hyperstimulation protocol was performed according to a long GnRH agonist protocol starting in the midluteal phase (day 21) of the preceding cycle. Embryos were assessed at 25 - 27 hr after ICSI for early cleavage. Embryos which reached the two cell stage at this interval were classified as Early Cleavage (EC) embryos, and the remaining as Non Early Cleavage (NEC) embryos. Embryos were assessed again at 64 - 68 hours post-ICSI for day-three embryo morphology. Day 3 embryo transfer was done. The best two or three embryos, according to day 3 embryo morphology were transferred. The patients were subdivided into two subgroups; one will transfer early cleavage embryos (EC) and the other will transfer non early cleavage embryo (NEC).

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 - 30 kg/m2
* Have two ovaries
* Regular cycles
* first ICSI cycle
* Long midluteal GnRH protocol.

Exclusion Criteria:

* uterine factor as a cause of female factor infertility
* pelvic masses or diseases (e.g: endometriosis, fibroids, hydrosalpnix, ...)
* history of medical disorders (e.g: hypertension, D.M, thyroid dysfunction, liver diseases, renal diseases,...)
* azoospermia as a cause of male factor infertility

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 193 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy | 6 weeks

SECONDARY OUTCOMES:
multiple pregnancy | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud edessy, prof, Study Director — Al-Azhar University; abd elnasr m ali, prof, Principal Investigator — Al-Azhar University; ahmed fata, prof, Principal Investigator — Al-Azhar University; wael hamed, dr, Study Chair — Al-Azhar University